CLINICAL TRIAL: NCT06529406
Title: Prospective Evaluation of Sequencing From antiCD-20 Therapies to Ozanimod (COAST: CD20 and Ozanimod Sequencing Trial)
Brief Title: Prospective Evaluation of Sequencing From antiCD-20 Therapies to Ozanimod
Acronym: COAST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1686
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — ozanimod

STUDY DESIGN:
Intervention Model Description: Ozanimod de-escalation of anti-CD20 treatment vs continued treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ozanimod de-escalation of anti-CD20 treatment (Experimental): Ozanimod will be started 6-12 months after the last anti-CD20 infusion, including ocrelizumab subcutaneous injection, or 30-180 days from their last ofatumumab injection. Ozanimod will be provided by the study.
  Interventions: Drug: Ozanimod
- Continued anti-CD20 treatment (No Intervention): Patients will continue to receive anti-CD20. Propensity score matched to the experimental arm.

INTERVENTIONS:
Drug: Ozanimod — De-escalation of anti-CD20 treatment using ozanimod.
  Other Names: Zeposia
  Arms: Ozanimod de-escalation of anti-CD20 treatment

SUMMARY:
A multi-center pilot study to evaluate safety and efficacy of ozanimod as de-escalation therapy in clinically stable MS patients previously treated with anti-CD20 therapy.

DETAILED DESCRIPTION:
Multicenter, Open Label, Prospective Study examining the safety and efficacy of de-escalation therapy to ozanimod (Zeposia®) over 36 months from anti-CD20 therapy for stable patients with relapsing forms of MS. A comparison to patients continuing anti-CD20 treatment was performed with propensity scoring to a cohort of at least 500 patients followed at Cleveland Clinic and the University of Colorado who also meet the above the inclusion and exclusion criteria. Patients were followed for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants have been diagnosed with relapsing forms of MS and have had multiple sclerosis related symptoms at least 3 years prior to baseline visit
* Male or female participants > or = to 18 years of age at the time of initiation of de-escalation
* Participants do not have evidence of new inflammatory disease activity (no new T2/contrast enhancing lesions, absence of relapses) for a minimum of two years prior to de-escalation
* Participant is taking an anti-CD20 therapy as a DMT continuously for a minimum of two years (e.g., has received at least 3 courses of rituximab, ocrelizumab, ublituximab; 24 months of treatment with ofatumumab; or a combination of treatments whereby the patient has been deemed to be B-cell depleted for 2 years) prior to initiation of de-escalation
* Participants received their last anti-CD20 infusion, including ocrelizumab subcutaneous injection, within 6-12 months or received their last ofatumumab injection within 30 -180 days from Day 1
* Participants must provide written informed consent and be able to comply with the visit schedule and study related assessments
* Participants must be able to undergo a brain MRI without anesthesia
* Woman of Childbearing Potential must agree to practice a highly effective method of contraception throughout the study until completion and willing to follow pregnancy precautions.

Exclusion Criteria:

* Any progression of neurological disability in the year prior to the screening visit that would be consistent with progressive MS
* Participant has an EDSS >6.5
* Participant has a history of other chronic neurological illnesses that might mimic MS with chronic or intermittent symptoms (i.e. ALS, myasthenia gravis, chronic neuropathy, etc.)
* Participant is considering pregnancy in the short term, is pregnant, lactating or has a positive serum beta human chorionic gonadotropin (B-hCG) measured during screening.
* Participant has any other significant medical or psychiatric illness, if uncontrolled, that could jeopardize a subject's health or put them at significant safety risk during the course of the study in the opinion of treating investigator. Examples: uncontrolled hypertension, uncontrolled diabetes, uncontrolled asthma, uncontrolled depression
* Participant has a history of cancer within the last 5 years, including solid tumors and hematological malignancies (except basal cell and in situ squamous cell carcinomas of the skin or cervical dysplasia/cancer that has been excised and resolved)
* Participant has a history in the last 6 months of myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, or Class III or IV heart failure
* Participant has Mobitz type II second-degree or third degree atrioventricular (AV) block, sick sinus syndrome, or sino-atrial block, unless the patient has a functioning pacemaker
* Participant has severe untreated sleep apnea
* Participant has a history of diabetes mellitus type 1, or uncontrolled diabetes mellitus type 2 with hemoglobin A1c (HbA1c) > 9%, or is a diabetic subject with significant comorbid conditions such as retinopathy or nephropathy, or a history of uveitis
* Participant has a history or known presence of recurrent or chronic infection (e.g., hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV); recurrent urinary tract infections are allowed.
* Any known or suspected active infection (excluding onychomycosis) at screening, including but not limited to a confirmed or suspected progressive multifocal leukoencephalopathy (PML). Known currently active tuberculosis (TB). History of incompletely treated Mycobacterium tuberculosis (TB) infection, as indicated by: Subject's medical records documenting incomplete treatment for Mycobacterium TB; Subject's self-reported history of incomplete treatment for Mycobacterium TB; Subjects with a history of TB who have undergone treatment accepted by the local health authorities (within 1 year from screening) may be eligible for study entry.

Exclusions related to Medications:

* Concomitant use of a monoamine oxidase inhibitor
* Use of systemic corticosteroids in the last 2 years, except for the use as a premedication for B-cell depleting treatment (Note: Use of inhaled or topical steroids; use of oral steroids for no greater than 14 days given for a non-MS condition are allowed)
* Prior use of alemtuzumab, mitoxantrone, cyclophosphamide, methotrexate, cyclosporine, or any experimental MS treatment within 5 half-lives
* Prior allergy to ozanimod

Exclusions related to Laboratory results:

* Participant has IgG levels <400 mg/dL
* Participant has neutrophils < 1500/μL (1.5 GI/L)
* Participant has an absolute white blood cell (WBC) count < 3500/μL (3.5 GI/L)
* Participant has an absolute lymphocyte count (ALC) < 800 cells/μL (0.80 GI/L).
* Participant has liver function impairment or persisting elevations of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) results > 3 x the upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
New T2 lesions count | 36 months
  Number of new T2 lesions on MRI scans.
Serious infections | 36 months
  Infections requiring hospitalization, intravenous antibiotic use, or prolonged antibiotic use for treatment of an infection for at least 30 days.

SECONDARY OUTCOMES:
Relapses | 36 months
  Protocol and/or suspected relapses
IgG and IgM levels | 36 months
  IgG and IgM levels
Infections | 36 months
  All infections including opportunistic infections.
No Evidence of Disease Activity (NEDA-3) | 36 months
  Not meeting any of the following criteria:
  1. Evidence of Relapse activity - collected every 3 months via phone calls/clinic visits.
  2. MRI disease activity - presence of new T2 lesions from MRI scans conducted at any timepoint.
  3. 6 months Confirmed Disability progression (CDP6): measured by the EDSS assessed at baseline and every 6 months. CDP6 is defined as an increase in Expanded Disability Status Scale (EDSS) score of ≥1.5 if baseline EDSS was 0; or ≥1.0 points if baseline EDSS was ≥0.5-≤5.5; or by ≥0.5 points if baseline EDSS ≥6, sustained over two consecutive visits.
Neurofilament light (NfL) and Glial Fibrillary Acid Protein (GFAP) | 36 months
  Neurofilament light (NfL) and Glial Fibrillary Acid Protein (GFAP)
Brain parenchymal and thalamic volume loss | 36 months
  Brain parenchymal and thalamic volume loss
Adverse Events | 36 months
  Adverse Events

OTHER OUTCOMES:
Symbol Digital Modalities Test | 36 months
  A 4 points or 10% change in cognition
9-hole peg test | 36 months
  A 20% change in hand function
25-foot walk speed | 36 months
  A 20% change in walking speed
Multiple Sclerosis Functional Composite (MSFC) | 36 months
  A change in any of the above three criteria
PRO outcomes | 36 months
  Include treatment satisfaction (TSQM), MS fatigue scale (Modified Fatigue Impact Scale [MFIS]), or quality of life (MSIS-29). A minimum of 5% change.
Changes in employment | 36 months.
  Changes in employment and full employment status.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Alvarez, MD/PhD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Cleveland Clinic, Las Vegas, Nevada
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with interest in multiple sclerosis. Data or samples shared will be coded with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement. For more information or to submit a request, please contact: clinicalresearchsupportcenter@ucdenver.edu

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT06529406/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT06529406/ICF_001.pdf